CLINICAL TRIAL: NCT04484454
Title: ProdromeNeuro: An Open-Label Study of Omega 3 Oil Nutritional Supplementation for Aging-Related Cognitive Decline
Brief Title: Open-Label Study of Omega 3 Oil Supplementation for Aging-Related Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: Prodrome Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProdromeNeuro
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Decline
Keywords: Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omega 3 Oil Supplementation (Experimental): Following all necessary screening, patients will be provided with the ProdromeNeuro Omega-3 oil supplement and instructed to consume the equivalent of 1 cc of the oil supplement per day for the first month, followed by 2 cc of the supplement/day for the second month, and finally ending with 4 cc/day of the supplement for the third month. Neurocognitive assessment and serology testing will take place at baseline, end of month 1, end of month 2, end of month 3, and one month post intervention-termination.
  Interventions: Dietary Supplement: ProdromeNeuro Omega 3 Oil Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: ProdromeNeuro Omega 3 Oil Nutritional Supplement — ProdromeNeuro is an algae-derived Omega 3 oil nutritional supplement product comprised of naturally occurring alkylglycerol and natural fatty acids. ProdromeNeuro functions as a natural plasmalogen precursor which can be administered orally.

SUMMARY:
Aging-related cognitive decline may be affected by brain cholesterol and the health of cell membranes. Certain nutritional supplements have been proposed to support membrane health, and there is increasing interest in plasmalogens and Omega-3 derived oil supplements to support brain health among older adults. The product being investigated in this study is the ProdromeNeuro Omega 3 oil nutritional supplement. This product contains naturally occurring fatty acids in higher concentrations than similar products that are commercially available. The purpose of this research study is to better understand the effects of ProdromeNeuro Omega-3 nutritional supplementation among subjects with age-related cognitive decline.

DETAILED DESCRIPTION:
There has been an increasing interest in plasmalogens as a potential therapeutic agent for age-related cognitive decline and neurodegenerative conditions, given the growing understanding of their involvement in key cellular functions as well as the clinical trends observed when plasmalogen levels are depleted. In addition to supporting the structural integrity of membranes, these plasmalogens are also involved in a variety of critically important cell functions: membrane fusion, ion transport, vesicle formation, and oxidation-reduction. Plasmalogen and serum plasmalogen deficiency has been shown to impair cellular functions, particularly related to cholesterol processing, and has been implicated in Alzheimer's and other diseases. Plasmalogen precursor supplementation has been demonstrated as safe and potentially efficacious in preclinical studies and some patient populations. In theory, ProdromeNeuro supplementation may yield therapeutic benefits among patients with age-related cognitive decline by increasing levels of neuroprotective plasmalogens.

The present study is being undertaken as an open-label study to evaluate the safety and tolerability of ProdromeNeuro Omega-3 Oil as an intervention for patients with age-related cognitive decline. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures. Neurocognitive assessment and serology testing kits to evaluate for plasmalogen levels will also be administered at baseline, end of the first month, end of the second month, end of the 3 month, and after one month post treatment termination.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive decline due to aging-related changes
* Clinical Dementia Rating stage of mild dementia 0.5 through moderate dementia CDR stages 1 and 2

Exclusion Criteria:

* Subjects unable to give informed consent
* Cognitive decline clearly related to an acute illness
* Subjects taking anticoagulants and anti-platelet agents
* Advanced terminal illness
* Any active cancer or chemotherapy
* Any other neoplastic illness or illness characterized by neovascularity

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Quick Dementia Rating Scale (QDRS) | Baseline
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
Montreal Cognitive Assessment (MoCA) | Baseline
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
30 Second Sit-Stand (30CST) | Baseline
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
Timed 25-foot Walk Test (T25FW) | Baseline
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
9 Hole Pegboard Task (9 HPT) | Baseline
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.

SECONDARY OUTCOMES:
QDRS | End of Month 1
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
QDRS | End of Month 2
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
QDRS | End of Month 3
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
QDRS | End of Month 4
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
MoCA | End of Month 1
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
MoCA | End of Month 2
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
MoCA | End of Month 3
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
MoCA | End of Month 4
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
30CST | End of Month 1
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
30CST | End of Month 2
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
30CST | End of Month 3
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
30CST | End of Month 4
  The 30-second chair stand involves recording the number of times that a person can complete a full stand in 30 seconds. This measure assesses functional lower extremity strength in older adults. The participant is instructed to complete as many full stands as possible within 30 seconds, starting in a seated position in the middle of an armless chair. The participant is instructed to fully sit between each stand. The tester silently counts the completion of each correct stand, and the score is the total number of stands within 30 seconds. The minimum clinically important difference (MCID) is 2 full stands per 30 second testing.
T25FW | End of Month 1
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
T25FW | End of Month 2
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
T25FW | End of Month 3
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
T25FW | End of Month 4
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25-foot walk. Scoring for this task is the average number of steps (from first step to the first heel-strike after the finish line) and time taken (seconds/milliseconds) of two trials. Minimally clinically important difference (MCID) is 20% improvement in time taken and/or number of steps taken to complete.
9HPT | End of Month 1
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
9HPT | End of Month 2
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
9HPT | End of Month 3
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
9HPT | End of Month 4
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

REFERENCES:
- [Background] Lee A, Gilbert RM. Epidemiology of Parkinson Disease. Neurol Clin. 2016 Nov;34(4):955-965. doi: 10.1016/j.ncl.2016.06.012. Epub 2016 Aug 18. PMID 27720003
- [Background] Trigiani LJ, Lacalle-Aurioles M, Bourourou M, Li L, Greenhalgh AD, Zarruk JG, David S, Fehlings MG, Hamel E. Benefits of physical exercise on cognition and glial white matter pathology in a mouse model of vascular cognitive impairment and dementia. Glia. 2020 Sep;68(9):1925-1940. doi: 10.1002/glia.23815. Epub 2020 Mar 10. PMID 32154952
- [Background] Dietschy JM, Turley SD. Cholesterol metabolism in the brain. Curr Opin Lipidol. 2001 Apr;12(2):105-12. doi: 10.1097/00041433-200104000-00003. PMID 11264981
- [Background] Mankidy R, Ahiahonu PW, Ma H, Jayasinghe D, Ritchie SA, Khan MA, Su-Myat KK, Wood PL, Goodenowe DB. Membrane plasmalogen composition and cellular cholesterol regulation: a structure activity study. Lipids Health Dis. 2010 Jun 14;9:62. doi: 10.1186/1476-511X-9-62. PMID 20546600
- [Background] Braverman NE, Moser AB. Functions of plasmalogen lipids in health and disease. Biochim Biophys Acta. 2012 Sep;1822(9):1442-52. doi: 10.1016/j.bbadis.2012.05.008. Epub 2012 May 22. PMID 22627108
- [Background] Muse ED, Jurevics H, Toews AD, Matsushima GK, Morell P. Parameters related to lipid metabolism as markers of myelination in mouse brain. J Neurochem. 2001 Jan;76(1):77-86. doi: 10.1046/j.1471-4159.2001.00015.x. PMID 11145980
- [Background] Rouser G, Yamamoto A. Curvilinear regression course of human brain lipid composition changes with age. Lipids. 1968 May;3(3):284-7. doi: 10.1007/BF02531202. No abstract available. PMID 17805871
- [Background] Engelmann B, Streich S, Schonthier UM, Richter WO, Duhm J. Changes of membrane phospholipid composition of human erythrocytes in hyperlipidemias. I. Increased phosphatidylcholine and reduced sphingomyelin in patients with elevated levels of triacylglycerol-rich lipoproteins. Biochim Biophys Acta. 1992 Nov 11;1165(1):32-7. doi: 10.1016/0005-2760(92)90072-4. PMID 1420345
- [Background] Mandel H, Sharf R, Berant M, Wanders RJ, Vreken P, Aviram M. Plasmalogen phospholipids are involved in HDL-mediated cholesterol efflux: insights from investigations with plasmalogen-deficient cells. Biochem Biophys Res Commun. 1998 Sep 18;250(2):369-73. doi: 10.1006/bbrc.1998.9321. PMID 9753636
- [Background] Poirier J, Miron J, Picard C, Gormley P, Theroux L, Breitner J, Dea D. Apolipoprotein E and lipid homeostasis in the etiology and treatment of sporadic Alzheimer's disease. Neurobiol Aging. 2014 Sep;35 Suppl 2(Suppl 2):S3-10. doi: 10.1016/j.neurobiolaging.2014.03.037. Epub 2014 May 15. PMID 24973118
- [Background] Leoni V, Solomon A, Kivipelto M. Links between ApoE, brain cholesterol metabolism, tau and amyloid beta-peptide in patients with cognitive impairment. Biochem Soc Trans. 2010 Aug;38(4):1021-5. doi: 10.1042/BST0381021. PMID 20658997
- [Background] Michikawa M, Fan QW, Isobe I, Yanagisawa K. Apolipoprotein E exhibits isoform-specific promotion of lipid efflux from astrocytes and neurons in culture. J Neurochem. 2000 Mar;74(3):1008-16. doi: 10.1046/j.1471-4159.2000.0741008.x. PMID 10693931
- [Background] Su XQ, Wang J, Sinclair AJ. Plasmalogens and Alzheimer's disease: a review. Lipids Health Dis. 2019 Apr 16;18(1):100. doi: 10.1186/s12944-019-1044-1. PMID 30992016
- [Background] Farooqui AA, Horrocks LA, Farooqui T. Glycerophospholipids in brain: their metabolism, incorporation into membranes, functions, and involvement in neurological disorders. Chem Phys Lipids. 2000 Jun;106(1):1-29. doi: 10.1016/s0009-3084(00)00128-6. PMID 10878232
- [Background] Zoeller RA, Lake AC, Nagan N, Gaposchkin DP, Legner MA, Lieberthal W. Plasmalogens as endogenous antioxidants: somatic cell mutants reveal the importance of the vinyl ether. Biochem J. 1999 Mar 15;338 ( Pt 3)(Pt 3):769-76. PMID 10051451
- [Background] Broniec A, Klosinski R, Pawlak A, Wrona-Krol M, Thompson D, Sarna T. Interactions of plasmalogens and their diacyl analogs with singlet oxygen in selected model systems. Free Radic Biol Med. 2011 Apr 1;50(7):892-8. doi: 10.1016/j.freeradbiomed.2011.01.002. Epub 2011 Jan 12. PMID 21236336
- [Background] Sindelar PJ, Guan Z, Dallner G, Ernster L. The protective role of plasmalogens in iron-induced lipid peroxidation. Free Radic Biol Med. 1999 Feb;26(3-4):318-24. doi: 10.1016/s0891-5849(98)00221-4. PMID 9895222
- [Background] Stables MJ, Gilroy DW. Old and new generation lipid mediators in acute inflammation and resolution. Prog Lipid Res. 2011 Jan;50(1):35-51. doi: 10.1016/j.plipres.2010.07.005. Epub 2010 Jul 23. PMID 20655950